CLINICAL TRIAL: NCT01900691
Title: Clinical Investigation to Evaluate Removal of the Evolution® Esophageal Stent - Fully Covered
Brief Title: Removal of the Evolution® Esophageal Stent - Fully Covered
Acronym: CLARITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-012
Record Dates: First submitted 2013-07-01; First posted 2013-07-16 (Estimated); Results first posted 2022-02-23 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Fistula; Esophageal Neoplasms; Esophageal Perforation; Esophageal Stenosis; Stents
Keywords: Esophageal Fistula; Esophageal Neoplasms; Esophageal Perforation; Esophageal Stenosis; Stents
MeSH Terms: conditions — Esophageal Fistula; Esophageal Neoplasms; Esophageal Perforation; Esophageal Stenosis

ARMS (1):
- Evolution® Esophageal Stent (Experimental)
  Interventions: Device: Evolution® Esophageal Stent - Fully Covered

INTERVENTIONS:
Device: Evolution® Esophageal Stent - Fully Covered — Placement of the Evolution® Esophageal Stent for benign or malignant strictures, fistulas, perforations or leaks with the intention of removal

SUMMARY:
The CLARITY study is a clinical trial approved by US FDA to study the removal of the Evolution® Esophageal Stent-Fully Covered in malignant and benign indications.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with benign or malignant stricture, fistula, perforation, or leak
* Physician plans to remove the stent within the duration of study follow-up

Exclusion Criteria:

* Patient is < 18 years of age
* Patient is unable or unwilling to provide written informed consent or comply with follow-up schedule
* Patient is pregnant, lactating, or planning on being pregnant within the next 6 months
* Patient is simultaneously participating in another investigational drug or device study
* Patient that is contraindicated to upper GI endoscopy and/or any procedure to be performed in conjunction with esophageal stent placement
* Patient has a known hypersensitivity or contraindication to study products that, in the opinion of the investigator, cannot be adequately pre-medicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-09; Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Vargo, M.D., M.P.H., Principal Investigator — The Cleveland Clinic
Locations (11):
- United States (11):
  - Mayo Clinic, Phoenix, Arizona
  - Harbor-University of California Los Angeles Medical Center, Torrance, California
  - Emory University Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Louisville, Division of Surgical Oncology, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Methodist Dallas Medical Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evolution® Esophageal Stent
Started | 130
Completed | 111
Not Completed | 19
Not completed — Death | 7
Not completed — Lost to Follow-up | 4
Not completed — Study Device Not Placed | 3
Not completed — Non study stent placed | 2
Not completed — Six month Follow up completed, stent not removed | 2
Not completed — Complete stent migration through digestive tract | 1

BASELINE CHARACTERISTICS:
Arm/Group | Evolution® Esophageal Stent
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Black | 11
  Ethnicity: Hispanic or Latino | 16
  Ethnicity: White | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Removal of Study Stent
Description: The study design allowed for 130 patients to be enrolled to ensure that 58 patients had an attempted endoscopic stent removal between 7 days and 6 months in order to assess the primary measure as per sample size calculation. Therefore, the first 58 patients (malignant or benign lesions) with data submitted regarding attempted endoscopic stent removal are included in this outcome measure. Successful stent removal is one in which the study stent is completely removed from the patient during a single endoscopic procedure with the wire mesh integrity maintained such that the stent can be removed in one contiguous piece. Additionally, successful stent removal includes no tissue damage or hemorrhage visible during the retrieval procedure that is both related to the endoscopic stent removal and requires immediate treatment.
Time Frame: 7 days to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Evolution® Esophageal Stent
Number analyzed (Participants) | 58
Participants | 57

2. Secondary Outcome: Number of Patients With Benign Indications That Achieved Clinical Success
Description: The rate of clinical success in patients with strictures that showed improvement or relief of dysphagia symptoms or a seal sufficient to enable oral intake in patients with fistulas, perforations, or leaks.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Evolution® Esophageal Stent: Evolution® Esophageal Stent - Fully Covered: Placement of the Evolution® Esophageal Stent for benign fistulas, perforations or leaks with the intention of removal
Arm/Group | Evolution® Esophageal Stent
Number analyzed (Participants) | 78
Participants | 44

ADVERSE EVENTS:
Time Frame: 6 months or removal of stent from patient (whichever comes first)
Arm/Group | Evolution® Esophageal Stent
All-Cause Mortality (participants affected / at risk) | 10/130
Serious Adverse Events (participants affected / at risk) | 46/130
Other Adverse Events (participants affected / at risk) | 94/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evolution® Esophageal Stent (N=130)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardic Arrythmia (Cardiac disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Retroperitoneal lymph adenopathy (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Erosive esophagitis (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Hematemesis (Gastrointestinal disorders) | 2 (2)
Intestinal ischemia (Gastrointestinal disorders) | 1 (1)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 7 (7)
Complication associated with device (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Sensation of foreign body (General disorders) | 4 (4)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Abdominal absces (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Fungemia (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7)
Sepsis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urossepsis (Infections and infestations) | 1 (1)
Pharyngeal prforation (Injury, poisoning and procedural complications) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Radiation pericarditis (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Esophageal adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Device dislocation (Product Issues) | 10 (10)
Confusional state (Psychiatric disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal compression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Central venous catheterization (Surgical and medical procedures) | 1 (1)
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evolution® Esophageal Stent (N=130)
Dysphagia (Gastrointestinal disorders) | 20 (20)
Device dislocation (Product Issues) | 84 (84)
Chest pain (General disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT01900691/Prot_SAP_001.pdf